CLINICAL TRIAL: NCT02009098
Title: Antibiotic Prophylaxis and Intervention for Postpartum Infections Following Caesarean Section
Brief Title: RCT of Postoperative Infections Following Caesarean Section Infections Following Caesarean Section
Acronym: APIPICS
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: Region of Southern Denmark (Other); University of Southern Denmark (Other); Hvidovre University Hospital (Other); Esbjerg Hospital - University Hospital of Southern Denmark (Other)
Responsible Party: Principal Investigator, Nana Hyldig, principal investigator, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2012-002068-29; 2012-002068-29 (EudraCT Number)
Record Dates: First submitted 2013-05-05; First posted 2013-12-11 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2014-10

CONDITIONS: Postoperative Infection
Keywords: Randomized Controlled Trial; Caesarean Section; preoperative; intraoperative; prophylactic antibiotics; antibiotics; timing; surgical site infections; endometritis; wound infections; urinary tract infections; infectious morbidity; neonatal antibiotics exposure; Antibiotic Prophylaxis
MeSH Terms: conditions — Surgical Wound Infection; Endometritis; Wound Infection; Urinary Tract Infections | interventions — Cefuroxime

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- præoperativ antibiotic (Active Comparator): iv Cefuroxime 1,5g administered 15-60 minutes before incision
  Interventions: Drug: Cefuroxime
- postoperativ antibiotic (Active Comparator): iv Cefuroxime 1,5g administered after umbilical cord clamping
  Interventions: Drug: Cefuroxime

INTERVENTIONS:
Drug: Cefuroxime — iv Cefuroxime 1,5g administered 15-60 minutes before incision versus iv Cefuroxime 1,5g administered after umbilical cord clamping
  Other Names: Cefuroxime "Fresenius Kabi"

SUMMARY:
Background Women undergoing Caesarean Section (CS) have an increased risk of postpartum infections compared to women undergoing vaginal delivery. In Denmark the incidence of post-CS infections is 7-10%. The most common infections are endometritis, Urinary tract infections (UTI) and wound infections (WI).

Prophylactic antibiotics are effective in preventing postoperative infections and national guidelines recommend that antibiotics should be administered as a single dose immediately before surgical incision. CS is an exception to this pre-incision administration approach. National guidelines recommend administration of antibiotics after umbilical cord clamping to avoid exposure of the child to antibiotics before birth. Recent studies of antibiotic prophylaxis for CS suggest that prophylactic antibiotics administered before incision compared to after umbilical cord clamping may reduce post-CS infections by up to 50%. Two Cochrane reviews from 2012 criticize these types of studies for lack of data for outcomes on the baby and on late infection in the mother.

This study is a double-blinded randomized controlled trial with a concurrent Health Economic Assessment. The study will examine the effect of change in timing of prophylactic antibiotics on the rate of post-CS infections (endometritis, UTI and WI). The study will be performed at the obstetric departments at Odense University Hospital (OUH), Hvidovre Hospital (HH) and Hospital South West Jutland (HSWJ) in collaboration with the Department of Clinical Microbiology, OUH, to ensure that the most appropriate antibiotic regime is used. Furthermore, collaboration with a neonatologist will ensure appropriate assessment of neonatal outcome.

The investigators plan to enroll the first patient at OUH February 2013. HH and HSWJ will follow with a couple of months delay. The inclusion period is scheduled to last until the investigators have 2844 participants, who have answered the questionnaire. The investigators expect to complete the inclusion period in October 2014 (last patient last visit, LPLV). Microbiological analyzes and data processing is expected to be completed one year after the LPLV. The study population is all women delivering a child by CS during the project period, at Department of Gynaecology and Obstetrics of OUH, HH and HSWJ.

Objective: Investigate whether and by how much antibiotics administered 15-60 minutes before incision versus after umbilical cord clamping reduces the rate of postpartum infections in a Danish population of women undergoing CS.

Hypothesis: Antibiotics administered pre-incision will result in fewer postoperative infections than antibiotics administered after the umbilical cord is cut.

Hypothesis: Antibiotics administered before incision are cost-effective, compared to administration after umbilical cord clamping, measured by post-CS infection and as cost per Quality Adjusted Life Year (QALY).

ELIGIBILITY:
All women delivering a child by CS at term, at Odense University Hospital, Hvidovre Hospital or Hospital of South West Jutland, Denmark, will be included in the study. Informed consent will be obtained during pregnancy.

Inclusion Criteria:

* Age ≥ 18 year
* Women, who can read and understand Danish
* A gestational age ≥ completed 28 weeks of gestation
* Rupture of membranes and active labour (uterine contractions) is allowed.

Exclusion Criteria:

* Hypersensitivity to cefuroxime or to any other cephalosporin antibiotics
* Previous immediate and/or severe hypersensitivity reaction to penicillin or any other beta-lactam antibiotic.
* Systemic exposure to any antibiotic agent within 1 week before delivery

  _ Antibiotic indicated due to PROM, fever or other indications at the time of caesarean section.
* Women being immunologically incompetent (e.g. HIV positive)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-10; Primary Completion 2015-10 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Women: The incidence of post-CS infection (endometritis, urinary tract infections, and wound infections) | within the first 30 days after surgery
  To be able to collect information about symptoms of infection after discharge a self-administered questionnaire will be sent to all participants within 30 days post-CS. Furthermore data on postoperative infections, recorded by diagnoses codes or surgical procedures, will be obtained from the Danish National Patient Registry.
Infant: admission to special care unit | participants will be followed for the duration of hospital stay, an expected average of 4 days

SECONDARY OUTCOMES:
Women: length of the primary and any secondary hospitalization | within the first 30 days after Caesarean Section
Women: readmissions to hospital/contact to the general practitioner on suspicion of infection after Caesarean Section | within the first 30 days after Caesarean Section
Women: antibiotic treatment on suspicion of infection after Caesarean Section | within the first 30 days after Caesarean Section
Infant: use of antifungal treatment against oral thrush | participants will be followed for the duration of hospital stay, an expected average of 4 days
Infant: necrotizing enterocolitis | participants will be followed for the duration of hospital stay, an expected average of 4 days
Infant: antibiotic treatment during hospital stay | participants will be followed for the duration of hospital stay, an expected average of 4 days
Infant: the need for intensive care treatment and length of stay in hospital | participants will be followed for the duration of hospital stay, an expected average of 4 days
Infant: Neonatal sepsis | participants will be followed for the duration of hospital stay, an expected average of 4 days
  Neonatal sepsis, Neonatal sepsis workup
Women: Number of Participants with Adverse Events as a Measure of Safety and Tolerability | participants will be followed for the duration of hospital stay, an expected average of 4 days
  Adverse reactions/events registered during hospitalization (complications, examinations, treatments, antibiotic use)

OTHER OUTCOMES:
Characteristics of the study population, which may affect the primary outcome "postoperative infections" | participants will be followed for the duration of hospital stay, an expected average of 4 days
  Date of admission, Date of birth, Birthplace, Date of discharges. Ethnicity, Maternal age, height and prepregnancy weight, Parity, Multiple gestations, Gravidity, Prior caesareans, Prior abdominal surgery, Drug/alcohol abuse, Diabetes mellitus, Preeclampsia, Smoking status, self-reported, Urine track infection (before birth). Presence of labor, Length of labor, Preterm labor, Rupture of membranes, Length of rupture of membranes, Number of vaginal examinations, Use of internal monitoring, Meconium, Use of antenatal steroids, cervical dilators, vacuum, amnioinfusion, extraamniotic saline infusion. Type of section, Anaesthesia type, Uterine incision type, Uterine closure layers, Uterine incision extensions, Need for transfusion, Intraoperative blood loss, Time of day, Operative time, Deviation from the standard surgical procedure. Birth weight (gram), Gestational age (week

CONTACTS AND LOCATIONS:
Overall Officials: Jan Stener Joergensen, MD, PhD, Study Chair — Odense University Hospital, department of Gynaecology and Obstetrics, University of Southern Denmark, Faculty of Health Sciences, institute of Clinical Research, research unit, department of Gynaecology and Obstetrics
Locations (3):
- Denmark (3):
  - Hospital of South West Jutland, Esbjerg
  - Hvidovre Hospital, Hvidovre
  - Odense University Hospital, Odense